CLINICAL TRIAL: NCT02106572
Title: Intravesical Mistletoe Extract in Superficial Bladder Cancer: A Phase III Efficacy Study
Brief Title: Therapeutic Instillation of Mistletoe
Acronym: TIM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abnoba Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB03; 2013-003446-16 (EudraCT Number); 2023-503718-66-00 (Other: EU CT No.)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2024-02

CONDITIONS: Superficial Bladder Cancer
Keywords: superficial bladder cancer; viscum album extract; mistletoe extract; abnobaVISCUM; recurrence rate
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — viscum album peptide; Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blind Review in accordance with with ICH-Biostatistics Guideline ICH E9
Oversight: Data Monitoring Committee: No

ARMS (2):
- abnobaVISCUM 900 (Experimental): intravesical instillation of abnobaVISCUM 900
  Interventions: Drug: abnobaVISCUM 900
- Mitomycin C (Active Comparator): intravesical instillation of Mitomycin C
  Interventions: Drug: Mitomycin C

INTERVENTIONS:
Drug: abnobaVISCUM 900 — intravesical instillation of abnobaVISCUM 900 13 times during treatment period
  Other Names: viscum album extract; mistletoe extract; abnobaVISCUM
  Arms: abnobaVISCUM 900
Drug: Mitomycin C — intravesical instillation of Mitomycin C 10 times during treatment period
  Other Names: MMC; Mitomycin
  Arms: Mitomycin C

SUMMARY:
The aim of this phase III study is to assess the efficacy of abnobaVISCUM® 900 compared with Mitomycin C (MMC) monotherapy in patients with superficial bladder carcinoma by evaluation of the time to tumor recurrence. Secondary objective is to evaluate the safety of abnobaVISCUM® 900, in particular, to compare the toxicity of the two treatments. Another secondary objective is the treatment efficacy as measured by calculated prognosis for recurrence and progression after 1 year, the tumor grading in case of a recurrence and by measurement of Quality of Life.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled, prospective, multinational Phase III confirmative study with 2 treatment groups and an adaptive design (Bauer and Köhne, 1994). The study is designed to compare the efficacy of treatment with abnobaVISCUM® 900 with Mitomycin C (MMC). Patients with completely resected superficial bladder carcinoma (Stage Ta) with an intermediate risk classification according to the European Association of Urology (EAU, update 2013) and with one immediately post operative MMC 40 mg or Epirubicin 50 mg intravesical instillation will be eligible for inclusion in the study.

The study comprises a screening period of not more than 6 weeks, a treatment period of 12 months for abnobaVISCUM® 900 and MMC and a follow-up period of 12 months. Patients will be screened within 6 weeks after the transurethral resection of the bladder (TURB) and the immediately post operative MMC 40 mg or Epirubicin 50 mg intravesical instillation. A re-resection should be performed before inclusion if indicated. Every patient is to provide written informed consent before any study related procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent for data protection and willingness to participate and comply with the study protocol prior to any study-related procedures
* Completely resected (detrusor muscle in the TUR specimen according to need) superficial bladder carcinoma (Stage Ta) with classification as intermediate-risk according to the EAU (update 2013) and one immediately post operative intravesical MMC 40 mg or Epirubicin 50 mg instillation, completed re-resection if indicated
* Karnofsky Performance Status of 50% to 100% (corresponding to Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2)
* Life expectancy of ≥ 2 years at the time point of study inclusion
* Normal renal and liver function, normal cardiac and hematology profiles (patients with laboratory values slightly outside the reference range may be included, unless the investigator considers the abnormality as clinically significant)
* Female patients of childbearing potential must have a negative pregnancy test (β-human chorionic gonadotropin test) at Screening. Pregnancy during the treatment period including 12 weeks after the last instillation has to be excluded

Exclusion Criteria:

* Locally infiltrative or metastatic bladder tumor (Stage T2 or greater), low-risk Ta tumor (primary, solitary, LG/G1, <3 cm, no CIS) or high-risk tumors according to EAU classification, update 2013 (T1; HG/G3; CIS; multiple and recurrent and large [>3 cm] Ta G1/G2 tumors [all conditions must be present at this point], presence of upper urinary tract tumors or lesions which were not completely removed by TURB
* Urinary tract infection, benign prostatic obstruction grade II or III, neurogenic bladder, stress incontinence, bladder or urethral diverticula, fistulas or urethral stenosis
* Patients with acute systemic illness, such as inflammatory infections with fever > 38°C
* Patients with previous recurrence of a superficial bladder cancer or radiotherapy of the bladder or other intravesical treatment within the last 6 months, or patients with previous mistletoe therapy
* Patients with other previous or co-existing malignancies or CIS
* Patients having any previous or concurrent therapy with a systemic chemo- / immunotherapeutical treatment regimen, in particular vinca alkaloids, bleomycine and doxorubicine, or patients who are treated with pyroxidine hydrochloride (vitamin B6)
* Untreated coagulation disorders or inadequate anticoagulation therapy
* Leukocyte count < 4,000/mm3 or platelet count < 100,000/mm3
* Serum creatinine > 1.7 mg/dL
* Patients with known hypersensitivity to the excipients of the study medication (monosodium phosphate, disodium phosphate, ascorbic acid)
* Patients with a known hypersensitivity to mistletoe products and MMC
* Patients who were administered within a 4-week period before Visit 1 any other experimental drug under investigation
* Male patients planning to father a child or sperm donation from the first administration of study medication until 3 months after the last administration of the study medication
* Male patients unwilling to use barrier contraception ie, condoms and spermicide, from the day of first administration of the study medication until 12 weeks after administration of the study medication. In case the sexual relation is restricted to women fulfilling one of the criteria listed under inclusion criteria for female patients the barrier contraception is not necessary.
* Patients with a history of alcohol and / or drug abuse
* Patients who are unable to be regularly observed, not permitting adequate follow-up and compliance to the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to tumor recurrence | up to two years
  The primary objective of the study is to assess the efficacy of abnobaVISCUM® 900. Primary efficacy criterion will be the time to tumor recurrence.

SECONDARY OUTCOMES:
Toxicity and tolerability of the study medication | up to two years
  The secondary objective, namely safety including toxicity and tolerability of the study medication, will be assessed by the monitoring of adverse events (AEs) according to the Common Terminology Criteria for Adverse Events (CTCAE), laboratory assessments (hematology, biochemistry and urinalysis) and a global judgment of tolerability.
Prognosis after 1 year for recurrence and progression | 1 year
  A secondary efficacy endpoint is prognosis after 1 year for recurrence and progression, estimated by the European Organization for Research and Treatment of Cancer (EORTC) Bladder Cancer Calculator.
Quality of Life with the EORTC QLQ-C30 and BLS24 Quality of Life Questionnaires | up to two years
  A secondary efficacy endpoint is measurement of Quality of Life with the EORTC QLQ-C30 and BLS24 questionnaires.
Tumor grading | up to two years
  A secondary efficacy endpoint is the tumor grading in case of a recurrence by cytology, ultrasound, and cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hess, Prof. Dr., Principal Investigator — Chief Medical Officer of the Urological Clinic of the University Hospital Essen
Locations (5):
- Theodor Bilharz Research Institute, Giza, Egypt
- Germany (4):
  - Clinic of Urology of the University Hospital of Essen, Essen
  - Urologische Gemeinschaftspraxis, Heinsberg
  - Urologische Praxis, Herzberg
  - Urologische Facharztpraxis, Würselen